CLINICAL TRIAL: NCT02750020
Title: Policy-Related Survey - Territory-wide Telephone Survey on Tobacco Control
Brief Title: Policy-related Survey on Tobacco Control
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Lam Tai-Hing, Sir Robert Kotewall Professor in Public Health, The University of Hong Kong
Other Study IDs: 2016 Policy Survey
Record Dates: First submitted 2016-04-13; First posted 2016-04-25 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Smoking
Keywords: Telephone survey
MeSH Terms: conditions — Smoking | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- never smokers: Around 1667 never smokers will be required to answer a questionnaire via telephone.
  Interventions: Other: Questionnaire
- ex-smokers: Around 1667 ex-smokers will be required to answer a questionnaire via telephone.
  Interventions: Other: Questionnaire
- current smokers: Around 1667 current smokers will be required to answer a questionnaire via telephone.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Current study is a retrospective telephone survey based on questionnaires. It aims to investigate the level of public support on current and future tobacco control measures and taxation policies and to address the timely impacts of smoke-free policies, substantiate public support on further tobacco control measures and assist COSH in shaping policy direction for government. The telephone survey will be conducted by a telephone survey agent under the monitor of applicants.

SUMMARY:
Current study is the fourth wave of the policy-related survey on tobacco control in Hong Kong. It aims to investigate the level of public support on current and future tobacco control measures and taxation policies and to address the timely impacts of smoke-free policies, substantiate public support on further tobacco control measures and assist COSH in shaping policy direction for government. In total, 5000 subjects will be randomly selected for a telephone interview. The subjects will be categorized into three groups, i.e. never smokers (1667), ex-smokers (1667) and current smokers (1667). They will be required to answer a questionnaire via telephone. All data shall be collected using a Computer Assisted Telephone Interview (CATI) system, which allows real-time data capture and consolidation. All interviews shall be conducted anonymously. Analysis of survey data will aim to identify current opinion on tobacco control policies and implications for future policies. Analyses will be controlled for confounding variables as required by stratification into sub-groups based on important pre-defined characteristics and/or by multivariate analysis. Comparison with past trends and, where possible, extrapolation of future trends will be explored. Weights will be applied to adjust for the sex and age of Hong Kong population, and to handle the over-sampling issues of current smokers. The data analysis will be conducted by statisticians.

DETAILED DESCRIPTION:
From 2013 to 2015, investigators conducted three waves of the policy-related survey on tobacco control. The surveys gathered information such as second hand smoking (SHS) exposure at home, in the workplace, and in various public places (e.g. bars/restaurants, door way of the buildings, streets, and bus stops), use of smoking cessation services, knowledge of smoking and quitting, and smoking prevalence; measured the impact of tobacco control policies such as tax increase in 2011 and 2014, expansion of smoke-free areas in 2009 and 2010, and pictorial health warnings on behavioral change of smokers and ex-smokers; collected the opinions on current policies such as smoke-free areas, pictorial health warnings and point of sale displays, and the opinions towards future policies such as tax increase, plain packaging, and tobacco endgame. The results of the three waves have been used by the Hong Kong Council On Smoking and Health (COSH) to advocate plain packaging, banning on point of sale displays, and increasing tobacco tax by 100% in the past 3 years.

In order to collect further information on issues related to tobacco control which should be addressed in future tobacco control measures in Hong Kong, COSH commissioned School of Public Health, HKU to conduct a fourth wave of the survey (2015/16). The current survey sought to use the Hong Kong data to update information on the prevalence of SHS and active smoking and its health effects, use of E-cigarettes, awareness of smoking cessation services and to identify the level of public support for current and future tobacco control measures as well as estimating the impact of existing policies.

ELIGIBILITY:
Inclusion Criteria:

* Aged 15 and above
* Cantonese speakers

Exclusion Criteria:

* Unable to provide a consent form
* Speak language other than Cantonese

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Hong Kong residents.
Sampling Method: Probability Sample
Enrollment: 5151 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Attitudes to tobacco control policies | Outcome will be assessed immediately after subjects answer the questionnaire as this is a cross-sectional survey.
  Telephone Survey

CONTACTS AND LOCATIONS:
Overall Officials: Tai Hing Lam, MD, Principal Investigator — School of Public Health, the University of Hong Kong
Locations (1):
- Public Opinion Programme, the University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No